CLINICAL TRIAL: NCT00564278
Title: Motivational Antidepressant Therapy for Hispanics
Brief Title: Effects of Adding Motivational Interviewing to Antidepressant Treatment for Hispanic Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Roberto Lewis-Fernandez, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #5516/#6609R; R01MH077226 (NIH); DSIR 82-SESC
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Depression
Keywords: Hispanic Americans; Major Depressive Disorder; Antidepressant Therapy; Motivational Interviewing; Treatment Retention; Treatment Adherence
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard antidepressant therapy (Active Comparator): Participants will receive standard antidepressant therapy, including selecting among 9 FDA-approved antidepressants from several classes.
  Interventions: Drug: Standard antidepressant therapy (SADT)
- Motivational antidepressant therapy (Experimental): Participants will receive motivational antidepressant therapy, including selecting among the same list of 9 FDA-approved antidepressants from several classes as in the control arm.
  Interventions: Drug: Standard antidepressant therapy (SADT); Behavioral: Motivational antidepressant therapy (MADT)

INTERVENTIONS:
Drug: Standard antidepressant therapy (SADT) — Treatment with medication will follow the Texas Medication Algorithm (TMA) for Depression. Antidepressant medications may include the following: citalopram (Celexa), escitalopram (Lexapro), paroxetine (Paxil CR), sertraline (Zoloft), venlafaxine XR (Effexor XR), bupropion SR (Wellbutrin SR), duloxetine (Cymbalta), nortriptyline (Pamelor), and mirtazapine (Remeron).
Behavioral: Motivational antidepressant therapy (MADT) — The same medication treatment for depression will be offered and supplemented with techniques from motivational interviewing.
  Arms: Motivational antidepressant therapy

SUMMARY:
This study will evaluate the effectiveness of adding motivational interviewing to antidepressant treatment for major depressive disorder in Hispanic adults.

DETAILED DESCRIPTION:
Depression is a serious illness that affects a person's mood, thoughts, and physical well-being. There are multiple types of depressive disorders, with major depressive disorder being one of the most common. The following symptoms may be signs of major depression: persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in previously enjoyed activities; excessive irritability and restlessness; suicidal thoughts; and inability to concentrate. Despite the widespread use of drug treatment for major depression in the United States, it continues to be underutilized in the Hispanic population. The retention rate in antidepressant therapy (ADT) among the Hispanic population is half that of the Caucasian population. It is believed that cultural factors and ambivalence toward seeking treatment interfere with ADT retention in Hispanic adults. Motivational antidepressant therapy (MADT) involves the use of motivational interviewing (MI) to discuss treatment with patients. This study will compare the effectiveness of culturally-specific MADT versus standard antidepressant therapy (SADT) in treating Hispanic adults with major depression.

Participants in this single-blind study will be randomly assigned to receive either MADT or SADT. A psychiatrist will conduct all medication visits and will recommend an initial antidepressant for each participant. Depending on treatment assignment, psychiatrists will use either the MADT or SADT approach in the medication visits. During the visits, participants will complete questionnaires, undergo vital sign measurements, and receive medication. Medication visits will occur weekly during the first two weeks, every 2 weeks for the next 6 weeks, and then on a monthly basis until the end of the study. In addition to visits with the psychiatrist, participants will complete 15-minute individual interviews with a clinician from the Hispanic Treatment Program. Individual interviews will take place every 2 weeks in the first month of treatment, monthly until the third month, and then every other month thereafter. The association between treatment, retention, and response will be assessed after 3 months of treatment. Preliminary outcome data will be obtained after 6 more months of continued treatment. After the end of treatment, participants may randomly be asked to participate in a small "focus group" to discuss personal experiences with study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Hispanic
* Meets Diagnostic and Statistical Manual, 4th edition criteria for major depressive disorder (MDD)
* Score of 16 or higher on Hamilton Depression Scale (HAM-D17) at study entry
* Willing to abstain from other psychotropic medications not included in the Texas Medication Algorithm (TMA) for depression, as clinically indicated, for the duration of the study. Zolpidem for insomnia will be allowed.
* Fluency in English or Spanish

Exclusion Criteria:

* Acute suicidality
* History of schizophrenia, bipolar affective disorder, schizoaffective disorder, depression with psychotic features, or organic brain syndromes
* Alcohol or other substance abuse or dependence (except nicotine) within 6 months prior to study entry
* Clinically unstable medical disease, including narrow-angle glaucoma or increased intra-ocular pressure
* Systemic blood pressure of 140/90 mm Hg or less
* Liver function test values two times above the normal level
* Pregnant or breastfeeding
* Sexually active women not using an effective method of birth control
* Current or past history of seizure disorder (except febrile seizure in childhood)
* Receiving effective medication for MDD
* Unable to tolerate or unwilling to accept drug-free period of varying length: 1 week for benzodiazepines taken as needed; 2 weeks for buspirone, lithium, anticonvulsants, stimulants, barbiturates, opiates, and regular-use benzodiazepines (except clonazepam); and 5 weeks for clonazepam
* Received electroconvulsive therapy (ECT) within 3 months prior to study entry
* Parkinson's disease, dementia of any type, or cognitive impairment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2008-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lewis-Fernandez, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vargas SM, Cabassa LJ, Nicasio A, De La Cruz AA, Jackson E, Rosario M, Guarnaccia PJ, Lewis-Fernandez R. Toward a cultural adaptation of pharmacotherapy: Latino views of depression and antidepressant therapy. Transcult Psychiatry. 2015 Apr;52(2):244-73. doi: 10.1177/1363461515574159. Epub 2015 Mar 3. PMID 25736422
- See also: Related info — https://nyculturalcompetence.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period extended from June 3, 2008 to Aug 14, 2013. Advertising was placed in local newspapers recruiting Hispanic adults to the trial, which took place in the Hispanic Treatment Program at the Psychiatric Institute, a research and clinical institute in Upper Manhattan affiliated with Columbia University.
Pre-assignment Details: Of N=109 patients enrolled in SADT, 12 were pre-treatment drops (signed consent but did not return for a medication visit) and N=97 came to 1+ medication visit. Of N=108 patients enrolled in MADT, 10 were pre-treatment drops (signed consent but did not return for a medication visit) and N=98 participated in at least one medication visit.
Groups:
- Standard Antidepressant Therapy: As per study criteria, the N=97 sample is our sample for data analysis. There were 37 men and 60 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline Hamilton Depression Scale-17 score of 16 or greater. Mean age was 43.41 (SD = 13.2).
- Motivational Antidepressant Therapy: As per study criteria, the N=98 sample is our sample for data analysis. There were 36 men and 62 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline Hamilton Depression Scale-17 score of 16 or greater. Mean age was 44.1 (SD = 12.3).
Period: Overall Study
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Started | 97 | 98
Completed | 50 | 56
Not Completed | 47 | 42
Not completed — Lost to Follow-up | 35 | 33
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 11 | 7

BASELINE CHARACTERISTICS:
Population: Patients who signed written informed consent and participated in baseline medication visit.
Groups:
- Standard Medication Therapy: N=97 patients were enrolled in this study arm and participated in at least one medication visit. There were 37 men and 60 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline HAMD-17 score of 16 or greater. Mean age was 43.4 with SD=13.2.
- Motivational Pharmacotherapy: N=98 patients were enrolled in this study arm and participated in at least one medication visit. There were 36 men and 62 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline HAMD-17 score of 16 or greater. Mean age was 44.1 with SD=12.3.
- Total: Total of all reporting groups
Arm/Group | Standard Medication Therapy | Motivational Pharmacotherapy | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 92 | 185
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.2) | 44.1 (12.3) | 43.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 98 | 195
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 97 | 98 | 195

OUTCOME MEASURES:

1. Primary Outcome: Number of Days in ADT (Retention)
Description: A continuous measure of the total number of days in treatment, based on visit attendance. At each kept visit, patients will be credited as having been in treatment for the number of days since their last scheduled visit. For example, patients attending sessions on weeks 0, 1, and 12 would have been in treatment for 35 days (7 [week 0 to week 1] + 28 [week 8 to week 12]).
Time Frame: Measured at Months 3 and 9
Population: Patients who signed consent and attended at least one medication visit.
Measure: Mean (Standard Deviation); unit: Days in treatment
Groups:
- Standard Antidepressant Therapy: N=97 patients were enrolled in this study arm and participated in at least one medication visit. There were 37 men and 60 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline HAMD-17 score of 16 or greater.
- Motivational Antidepressant Therapy: N=98 patients were enrolled in this study arm and participated in at least one medication visit. There were 36 men and 62 women. All were of Hispanic ethnicity, as the study focused on this population exclusively. All were depressed, with a baseline HAMD-17 score of 16 or greater.
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
Days in treatment
  Days in txt at 3 months | 59.5 (30.65) | 65.5 (24.6)
  Days in txt at 9 months | 148.7 (99.3) | 164.1 (89.2)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; We also conducted an analysis using a Generalized Estimating Equations model adjusting for a number of covariates. We will conduct a three-part regression analysis assessing early/middle/late effects of MPT on retention. We will also conduct moderator analyses, as described in the original study grant, to determine whether there are specific patient groups for whom a significant difference in days in treatment is found; Test type: Superiority or Other; p = 0.26, t-test, 2 sided — All analyses presented are at 9 months; t(193) = -1.14, p=.26; GEE model Beta = 17.46, 95% CI 2-sided [-16.61 to 51.53]

2. Primary Outcome: Mean of Depressive Symptoms Over 36-week Follow-up Using Hamilton Depression Scale -17-item Version (Symptoms)
Description: Depressive symptoms were assessed using the 17-item standard clinician-administered version of the Hamilton Depression Scale (HAMD-17). We analyzed the HAMD-17 score, calculated as the sum of the individual items and ranging from 0 to 35 with higher numbers indicating more symptoms. HAMD-17 was assessed at baseline and the follow-up visits specified below.
  We calculated the model-estimated mean of the HAMD-17 over 36 weeks using repeated measures.
Time Frame: HAMD-17 assessed at follow-up weeks 2, 4, 8, 12, 20, 28, and 36.
Population: All patients enrolled in both arms with available data at assessment time points.
Measure: Mean (Standard Deviation); unit: units on a scale ranging from 0 to 35
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
units on a scale ranging from 0 to 35 | 12.08 (7.17) | 11.71 (7.31)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See Method of Estimation below; Mixed Model Beta for MADT vs SADT = -0.28, 95% CI 2-sided [-1.57 to 1.01] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline depressive symptoms and time to assess the effect of MADT vs. SADT on mean depressive symptoms over follow-up

3. Primary Outcome: Mean Disability Over 36-week Follow-up Using Sheehan Disability Scale (Impairment)
Description: Psychosocial functioning was assessed using the Sheehan Disability Scale (SDS), a self-report instrument composed of three visual analog subscales assessing degree of disruption caused by symptoms in three domains: work, social/leisure activities, and family/home life. We analyzed the 3 subscale scores for the 3 domains separately which ranged from 0 to 10 with higher scores indicating worse functioning. The SDS was assessed at baseline and the follow-up visits specified below. We calculated the model-estimated mean of the SDS over 36 weeks using repeated measures.
Time Frame: SDS at follow-up weeks 2, 4, 8, 12, 20, 28, and 36.
Population: Patients with available data at assessment time points.
Measure: Mean (Standard Deviation); unit: Units on a scale ranging from 0-10
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
Units on a scale ranging from 0-10
  Work | 4.36 (3.44) | 4.93 (3.41)
  Social/leisure | 4.87 (3.29) | 5.44 (3.27)
  Family/home life | 4.55 (3.14) | 5.05 (3.23)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See under Method of Estimation, below; Work - Mixed Model Beta for MADT vs SADT = 0.22, 95% CI 2-sided [-0.50 to 0.95] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline work-related disability score and time to assess the effect of MADT vs. SADT on mean disability score in the work domain over follow-up
Statistical Analysis 2: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See under Method of Estimation below; Social-Mixed Model Beta for MADT vs SADT = 0.22, 95% CI 2-sided [-0.49 to 0.92] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline social-related disability score and time to assess the effect of MADT vs. SADT on mean disability score in the social domain over follow-up
Statistical Analysis 3: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See Method of Estimation below; Family-Mixed Model Beta for MADT vs SADT = 0.55, 95% CI 2-sided [-0.08 to 1.18] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline family-related disability score and time to assess the effect of MADT vs. SADT on mean disability score in the family domain over follow-up

4. Primary Outcome: Mean Perceived Quality of Life Over 36-week Follow-up Using Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)
Description: Quality of life was assessed using the 16-item Short Form of the Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ), a self-reported measure of quality of life in 8 domains that is sensitive to depressive symptom severity and treatment response. We analyzed the QLESQ total score as a percentage of the maximum possible score (ranging from 0-100) to facilitate comparisons across areas of functioning. It was calculated as such: % Max = (Raw score - minimum possible score) / (maximum possible score-minimum possible score) where raw score is the sum of the first 14 items. Higher numbers indicate better quality of life, greater enjoyment, and satisfaction. The QLESQ was assessed at baseline and the follow-up visits specified below. We calculated the model-estimated mean of the QLESQ over 36 weeks using repeated measures.
Time Frame: QLESQ at follow-up weeks 2, 4, 8, 12, 20, 28, and 36.
Population: Patients with available data at assessment time points.
Measure: Mean (Standard Deviation); unit: percentage of maximum possible score
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
percentage of maximum possible score | 50.05 (18.59) | 48.92 (19.50)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See Method of Estimation, below; Mixed Model Beta for MADT vs SADT = 0.02, 95% CI 2-sided [-3.61 to 3.64] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline QOL score and time to assess the effect of MADT vs. SADT on mean percent of quality of life over follow-up

5. Secondary Outcome: Mean Patient Satisfaction Over 36-week Follow-up Using Client Satisfaction Questionnaire (CSQ)
Description: Patient satisfaction was assessed using the 8-item Client Satisfaction Questionnaire (CSQ) which assesses patients' satisfaction with the services received. CSQ total score ranges from 8-32 with higher scores indicating greater satisfaction. The CSQ was assessed at baseline and the follow-up visits specified below. We calculated the model-estimated mean of the CSQ over 36 weeks using repeated measures.
Time Frame: CSQ at follow-up weeks 2, 4, 8, 12, 20, 28, and 36.
Population: Patients with available data at assessment time points.
Measure: Mean (Standard Deviation); unit: units on a scale ranging from 8 to 32
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
units on a scale ranging from 8 to 32 | 27.59 (3.38) | 27.41 (3.39)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See Method of Estimation below; Mixed Model Beta for MADT vs SADT = -0.04, 95% CI 2-sided [-0.74 to 0.66] — A Generalized Linear Mixed Model was used with random intercept for clinician adjusted for baseline patient satisfaction and time to assess the effect of MADT vs. SADT on mean patient satisfaction over follow-up

6. Secondary Outcome: Proportion of Fully Adherent Days
Description: We used the Composite Adherence Score (CAS) described in our grant application to calculate medication adherence levels from all data sources (electronic caps [eCaps], pill count, self-report) and compare these across arms. Calculated via a statistically calibrated algorithm, the CAS relied first on eCaps data, secondarily on pill count, and the adherence questionnaire if eCaps data was missing due to an eCap malfunction. We calculated the number of the days the patient was fully adherent, number of days of partial adherence (e.g., opened the eCap fewer times than prescribed), or number of days of nonadherence when they did not take any prescribed pills. Patients who dropped out of the study and provided no further follow-up data were considered nonadherent for the remainder of the study period. We calculated the therapy-adherent period as a proportion of the total intended treatment period or proportion of days of full adherence, # of fully adherent days / # of days in treatment.
Time Frame: Measured at each visit, up to 36 weeks
Population: All patients in both arms
Measure: Mean (Standard Deviation); unit: Proportion of Fully Adherent days
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Number analyzed (Participants) | 97 | 98
Proportion of Fully Adherent days | 0.47 (0.34) | 0.56 (0.32)
Statistical Analysis 1: Comparison: Standard Antidepressant Therapy vs Motivational Antidepressant Therapy; Test type: Superiority or Other; See Method of Estimation below; Mixed Model Beta for MADT vs SADT = 9.14, 95% CI 2-sided [2.71 to 15.57] — A Generalized Linear Mixed Model was used with random intercept for clinician to model the effect of MPT vs. SADT on the mean proportion of fully adherent days over the study period. We used an exchangeable covariance structure

ADVERSE EVENTS:
Time Frame: Time frame was duration of study: maximum of 36 weeks.
Groups:
- Standard Antidepressant Therapy: Participants will receive standard antidepressant therapy. Standard antidepressant therapy (SADT): Treatment with medication will follow the Texas Medication Algorithm (TMA) for Depression. Antidepressant medications may include the following: citalopram (Celexa), escitalopram (Lexapro), paroxetine (Paxil CR), sertraline (Zoloft), venlafaxine XR (Effexor XR), bupropion SR (Wellbutrin SR), duloxetine (Cymbalta), nortriptyline (Pamelor), and mirtazapine (Remeron).
- Motivational Antidepressant Therapy: Participants will receive motivational antidepressant therapy. Motivational antidepressant therapy (MADT): The same medication treatment for depression will be offered as in the SADT arm and supplemented with techniques from motivational interviewing.
Arm/Group | Standard Antidepressant Therapy | Motivational Antidepressant Therapy
Serious Adverse Events (participants affected / at risk) | 1/97 | 2/98
Other Adverse Events (participants affected / at risk) | 3/97 | 5/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Antidepressant Therapy (N=97) | Motivational Antidepressant Therapy (N=98)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Pt developed suicidal ideation during trial. After phone eval, he was referred to psych ER, from where he was admitted to inpatient psychiatric unit. After discharge, pt requested study termination and follow-up in non-research outpatient unit.
Manic episode (Psychiatric disorders) | 0 (0) | 2 (2) — Pt without clear history of bipolar disorder developed manic episode when started on antidepressant. Antidepressant was discontinued and appropriate mood stabilizers were initiated. Pt was terminated from the study and treated openly.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Antidepressant Therapy (N=97) | Motivational Antidepressant Therapy (N=98)
Neck stiffness or soreness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
Focused only on Hispanics, so applicability to other populations unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No